CLINICAL TRIAL: NCT00351481
Title: Recurrent Embryo Implantation Failure in Women Undergoing IVF/ ICSI; an Investigation of the Intra-Uterine Environment During the Window of Implantation
Brief Title: Failure of Implantation After Recurrent Embryo Transfers
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Other Study IDs: FIRE-study
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2007-04

CONDITIONS: Infertility
Keywords: IVF; endometrial receptivity; embryo implantation; recurrent implantation failure
MeSH Terms: conditions — Infertility

SUMMARY:
We will investigate maternal and embryonic factors in women with recurrent implantation failure, undergoing IVF/ ICSI treatment. Women who have not achieved a pregnancy after three embryo transfer procedures will undergo an endometrial biopsy during the window of implantation in a natural cycle. During the next treatment cycle we will aspirate endometrial secretion and perform a doppler ultrasound investigation of the a. uterina. Moreover, we will investigate the cytokine expression from the transferred embryo from the culture medium.

DETAILED DESCRIPTION:
Rationale:

Despite advances in IVF procedures and the transfer of embryos of high morphological quality embryos, pregnancy rates from IVF remain around 30% per embryo transfer procedure. Failure of the transferred embryo to implant remains the most important limiting factor determining in vitro fertilization (IVF) or intra cytoplasmic sperm injection (ICSI) success rates. If progress is to be made in improving implantation rates, a greater understanding of the factors which determine successful implantation is required. Recurrent implantation failure after IVF may be due to an endometrial, and embryo problem or both. All women entering our IVF program undergo pre-conceptional counseling and a pre-treatment blood withdrawal for hormonal investigation and investigation of uterine cavity by ultrasound examination, hysteroscopy and endometrial biopsy. The data generated by this pre-treatment screening potentially enables factors predictive of implantation failure to be identified. In addition, study of the further IVF cycle will increase our knowledge of the factors of endometrial and embryo factors involved in implantation failure, and aid in the characterization of the different causes of this distressing clinical problem. On the basis of these data, rational interventions designed to improve outcome can be designed and tested.

Objective:

To delineate pre-treatment predictors of recurrent implantation failure, to characterize the different phenotypes of women suffering from this problem and to study the relative importance of maternal and embryonic causes of implantation failure.

Study design:

Prospective, controlled cohort study.

Study population:

50 women who have received at least 3 embryo transfers in previous IVF cycles carried out within the UMC Utrecht, without achieving a clinical pregnancy. The control group of 'normal implanters' consists of 30 women who have previously readily conceived following ICSI for the treatment of severe male subfertility.

Main study parameters/endpoints:

1. Retrospective analysis of screening parameters, including analysis of endometrial biopsy material for Noyes criteria of endometrial dating, uterine natural killer (uNK) cell count and dietary/ lifestyle parameters obtained by questionnaire during pre-conceptional counseling.
2. Analysis of uNK cell count obtained from luteal phase endometrial biopsy prior to the treatment cycle.
3. Analysis of endometrial secretion and embryo culture medium cytokine expression profile measured at the time of embryo transfer in a subsequent IVF cycle: comparison with normal profile identified in the ICE study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Much of the data to be analysed will be collected from routine clinical work up (pre-conceptional screening). Women with recurrent implantation failure then embarking on a further IVF cycle will be invited to participate in this study and will undergo additional investigation. This will include an endometrial biopsy prior to the treatment cycle, and endometrial fluid aspiration prior to embryo transfer in the subsequent treatment cycle. No negative effect on pregnancy rates from these interventions have been reported. The theoretical risk associated with the aspiration of endometrial secretion before embryo transfer might be disruption of embryo implantation. However, our group has developed a technique which, as we have previously shown, does not disrupt the process of implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women who have not achieved a pregnancy, despite 3 subsequent embryo transfers, of which only one is allowed to be a transfer of a cryo-thawed embryo. A chemical pregnancy or E.U.G. will not be regarded as a pregnancy. An abortion will be regarded as a pregnancy.

Exclusion Criteria:

* women older than 37 years.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Macklon, Professor, Study Chair — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] van der Gaast MH, Beier-Hellwig K, Fauser BC, Beier HM, Macklon NS. Endometrial secretion aspiration prior to embryo transfer does not reduce implantation rates. Reprod Biomed Online. 2003 Jul-Aug;7(1):105-9. doi: 10.1016/s1472-6483(10)61737-3. PMID 12930588